CLINICAL TRIAL: NCT04426123
Title: Masseter Myofascial Pain Relief Following an Intra-muscular Injection With Botulinum Toxin Type A: A Randomized Double-blind Controlled Multicenter Pilot Study
Brief Title: Masseter Myofascial Pain Relief Following an Intra-muscular Injection With Botulinum Toxin Type A.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Region Örebro County (Other)
Collaborators: Region Västmanland (Other); Landstinget i Värmland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 273697
Record Dates: First submitted 2020-05-29; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-04

CONDITIONS: Myalgia; Myofascial Pain
MeSH Terms: conditions — Myalgia | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin (Active Comparator): Botulinum toxin type A
  Interventions: Drug: Botulinum toxin type A
- Saline solution (Placebo Comparator): NaCl
  Interventions: Other: saline solution

INTERVENTIONS:
Drug: Botulinum toxin type A — Intramuscular injection with Botulinum toxin type A in m.masseter and m.temporalis.
  Other Names: Botox
  Arms: Botulinum toxin
Other: saline solution — Intramuscular injection with NaCl in m.masseter and m.temporalis.
  Other Names: Physiologic NaCl
  Arms: Saline solution

SUMMARY:
Investigating the effect of a single intramuscular injection with botulinum toxin (BTX) compared to NaCl in patients with jaw muscle myalgia.

This investigation is designed as an double blind multicenter pilot study for hypothesis generation on 48 patients with chronic jaw muscle myalgia at four specialist dental clinics. The subjects visit the clinic on 3 predefined occasions, one telephone call and one scheduled evaluation by mail.

The objective is primarily to evaluate the change in number of days with pain at two months following one session of BTX injections of the masseter and temporalis muscles in subjects with jaw muscle myalgia pain.

The outcome of this study will serve as a basis for a later randomized controlled trial

DETAILED DESCRIPTION:
Temporomandibular disorders (TMD) is the second most common musculoskeletal condition (after chronic low back pain) and refer to pain and dysfunction in the temporomandibular system and its muscles, joints, and associated structures. The prevalence of TMD is 4-15% among adults where myalgia is the most common form of TMD.

Diagnostic Criteria for temporomandibular disorders (DC/TMD) was introduced in 2014 and is used worldwide for classifying TMD. Myalgia is the second group of disorders of DC/TMD and is defined by pain in a masticatory structure that is modified by jaw movement, function, or parafunction and familiar pain in masticatory muscle(s) with either muscle palpation or maximum opening.

Myofacial pain is the most common form of TMD, affecting about half of the patients presenting in TMD clinics. Myofascial pain is usually treated with conservative treatment including occlusal, physical and pharmacologic therapies. However, there is no evidence on which conservative treatment is the most beneficial in treating myalgia pain, mainly due to lack of randomized controlled trials.

Botulinum toxin A (BTX) is a neurotoxin isolated from Clostridium botulinum. Injected into a muscle the effect occurs in the presynaptic junction by blocking the release of acetylcholine, resulting in weakening of the muscular activity by affecting alpha and gamma motor neurons. The clinical effect occurs after 3-7 days after administration with a duration of up to 4 months. The BTX-effect diminish when new formation of synaptic connections occur due to sprouting.

Regional myofascial pain is characterized by the presence of trigger points and BTX, as a potent neurotoxin, has been used for its treatment. However, a Cochrane review reported inconclusive evidence to support the use of BTX in the treatment of myofascial pain. In another Cochrane review on cervical dystonia significant improvements were found with odds ratio (OR) of 20% in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) total score after four weeks (OR 4.69; 95% CI 2.06 to 10.69) and a weighted mean difference of -5.92 (95% CI -9.61 to -2.23). Studies investigating the effect of BTX on masticatory muscle myalgia have been summarized in systematic reviews and with inconclusive evidence to support the effect of BTX. Meta-analyses were inconclusive due to the heterogeneity of the studies and methodological flaws.

There are several theories of how BTX may reduce myalgia. Assuming myalgia is caused by muscle hyperactivity, BTX will reduce hyperactivity and thereby pain. In the presence of trigger points within the muscle, BTX may eliminate the triggers and then reduce pain. In case of muscle inflammatory pain, BTX reduces muscle activity and may then facilitate reduction of inflammation and consequently the pain. This can be caused by blocking the release of neurotransmitters such as substance P and glutamate. In conclusion, the mechanism on how muscle paralysis reduces pain is not clear.

A drawback of BTX-treatment is the potential side effects not found for other treatments of myalgia pain. Minor complications associated with any intra-muscular injection are pain, bruising and swelling. Some patients develop severe headache, muscle atrophy and paralysis in areas adjacent to the injection site causing ptos, difficulty in speaking, swallowing and respiratory problems. The risk-benefit relation is not established when treating masticatory myalgia.

The National Board of Health and Welfare in Sweden does not recommend the use of BTX for treating myofascial pain because of insufficient scientific evidence. The key publications on BTX for the treatment of jaw muscle pain are using reduction of pain intensity as the primary measure which may be a blunt parameter to evaluate treatment effects of chronic pain.

Therefore, there is a need to explore BTX-treatment effects of jaw muscle myalgia in relation to side effects using a set of measures to be used for hypothesis generation.

The purpose of this study is to help fill one of the knowledge gaps and be a valuable addition to increasing the quality of treatments made on the group of people diagnosed with myalgia in the masticatory system.

This study is targeted to include a total of 48 subjects with the diagnosis myalgia. Half of the subjects will receive one injection of botulinum toxin type A in their masseter and temporalis muscles. The other half will be the placebo group receiving NaCl injection on the same sites.

Injection treatment is made bilaterally independent of the presence of bilateral or unilateral myalgia.

A randomization list is generated by computer and each randomization should be balanced with as many subjects in the treatment group as in the control group. Randomization will be made in blocks of four. The randomization, which is sealed in individual envelopes, is performed by a person who is not attached to the project and keeps the randomization list locked up. The envelopes contain the randomization number and description of the substance to be injected. The envelope is opened immediately before the treatment and after all inclusion criteria and exclusion criteria are met.

After the investigator has checked alignment to the inclusion/exclusion criteria the study nurse will prepare the syringes in a separate room according to the randomization envelope information. The opened randomization envelope will then be put in a larger envelope which will be sealed and stored in the CRF-binder. The syringes will then be provided to the investigator without her/his knowledge on its content.

A paper-based Case Report Form (CRF) is used for data collection. The investigator must ensure that data is registered and any corrections in the CRF are made as stated in the study protocol and in accordance with the instructions.

The study team at each center consists of a dentist and a study nurse. The subjects visit the clinic on 3 predefined occasions, one telephone call and one scheduled evaluation by mail.

Visit 1: Enrollment, subject information and informed consent. After checking the inclusion and exclusion criteria the subject is assigned an enrollment number. Clinical examination is performed by the dentist. Questionnaires and diaries are handed out and the patient is instructed.

Visit 2: This visit will be done 2 weeks after enrollment visit. A baseline clinical examination is done. Questionnaires and diary are returned. After checking the inclusion and exclusion criteria the intervention substance is prepared according to the randomization code and the dentist performs the injection treatment. The subject is instructed how to complete a new set of questionnaires. Adverse events are registered.

By mail evaluation: Two weeks (+ 4 days) after visit 2. The patient returns the questionnaires and diaries by surface-mail.

Telephone evaluation: One month (+ 1 week) after visit 2. Telephone call. Adverse events are registered.

Visit 3: Two months (+ 2 weeks) after visit 2. The dentist collects questionnaires and diaries and a clinical examination is made. The subject is then completed within the scope of the study. Adverse events are registered. If further treatment is required, it is made outside the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* > 3-month complaints of jaw/face pain
* the diagnose myalgia according to DC/TMD
* understands Swedish verbally and in writing
* in writing give his/her consent to participate

Exclusion Criteria:

* polyarthritis/connective tissue disease
* fibromyalgia or other generalized pain
* neurological disorders
* whiplash associated disorders
* ongoing virus or bacterial infection
* ongoing dental treatment
* botulinum toxin injection in the jaw or face past six months
* complex psychiatric/psychological profile, institutional residence
* employee at the trial clinic, internal resident
* hypersensitivity to botulinum toxin, human albumin
* serious health conditions according to the examiner's assessment
* in the presence of infection at the proposed injection site(s)
* pregnancy or lactating
* fertile women not on contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain days | 2 months
  The change in frequency (number) of pain days

SECONDARY OUTCOMES:
Pain intensity | 2 months
  Change in average pain intensity by answering the question: "In the past two weeks", on the average, how intense was your pain rated on a 0-10 scale where 0 is "no pain" and 10 "pain as bad as could be" (That is, your usual jaw pain at times you were experiencing pain)".
Pain intensity on maximal opening of the jaw | 2 months
  Change of pain intensity at maximal opening of the jaw. The subject will assess their jaw pain on maximal opening on a numeric rating scale 0-10, where 0 is no pain and 10 is worst pain imaginable.
JFLS-20 | 2 months
  Change in physical function: Jaw functional problems will be evaluated using the 20-item global Jaw Functional Limitation Scale (JFLS-20), with possible mean scores ranging from 0-10, where 0 i no limitation and 10 is severe limitation.
PHQ-9 | 2 months
  Change in emotional function using the Patient Health Questionnaire-9 (PHQ-9), a multipurpose instrument used for screening, diagnosing and measuring depression severity, with possible scores ranging from 0-27, where higher scores indicate more severity.
PGIC | 2 months
  Global improvement. At the follow-up visit the subjects will rate the change in their overall status since beginning the study treatment using the Patient Global Impression of Change (PGIC) scale, a 7-point scaled instrument ranging from "very much improved" to "very much worse"
GCPS | 2 months
  Change in the Graded Chronic Pain Scale, GCPS, pain and its consequences. GCPS assesses 2 dimensions of overall chronic pain severity: pain intensity and pain-related disability. For pain intensity a numeric rating scale 0-10 is used, where 0 is no pain and 10 is worst pain imaginable. For pain-related disability a numeric rating scale from 0-10 is used where 0 is 'no interference' and 10 is 'extreme change'.

CONTACTS AND LOCATIONS:
Overall Officials: Göran Isacsson, Assoc. Prof., Study Director — Region Stockholm; Mohamad Schumann, DDS, Study Director — Västerås; Daniel Ovesson, DDS, Study Director — Karlstad

IPD SHARING:
Plan to Share IPD: No